CLINICAL TRIAL: NCT02234596
Title: Phase II Trial of Nintedanib in Patients With Advanced Esophagogastric Cancer
Brief Title: Nintedanib in Patients With Advanced Esophagogastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-094
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Results first posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2020-04

CONDITIONS: Esophagogastric Adenocarcinoma
Keywords: Nintedanib; 14-094
MeSH Terms: interventions — nintedanib

ARMS (1):
- Nintedanib (Experimental)
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — Nintedanib 200mg twice daily administered continuously. Patients will continue on treatment until progression of disease. Each cycle consists of 28 days continuously, unless interrupted for intolerable toxicity.

SUMMARY:
This is a phase II study of Nintedanib in patients with metastatic or recurrent esophagogastric cancer. The goal of the study is to evaluate the efficacy of Nintedanib, an orally available triple kinase inhibitor targeting the receptors of the vascular endothelial growth factor (VEGF), platelet derived growth factor (PDGF), and fibroblast growth factor (FGF) receptor pathways.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically MSKCC confirmed esophagogastric adenocarcinoma.
* Metastatic diseases measurable or evaluable on a CT or MRI scan according to RECIST 1.1 criteria. Locally recurrent disease that is not amenable to potentially curative surgery or radiation therapy is also allowed. Lesions must be ≥10mm in size. Recurrent or metastatic disease within a prior radiation field is acceptable as long as the disease has progressed in the radiation field by RECIST criteria.
* Patients are allowed to have had a maximum of 1 prior chemotherapy regimen for metastatic disease. Patients are allowed to have a maximum of two prior regimens if they previously received neoadjuvant/adjuvant chemotherapy or chemoradiotherapy for their initial localized disease.
* Patients aged 18 years or older.
* Life expectancy of at least 6 months.
* Karnofsky Performance Status (KPS) performance score ≥ 70%.
* Patients must be able to reliably take and swallow oral medications.
* Patients with prior deep vein thrombosis (DVT) or pulmonary embolism (PE) currently on anticoagulation regimen will be permitted.
* Adequate bone marrow, liver, and renal function as assessed by the following:
* Hemoglobin ≥ 9.0 g/dL.
* Absolute neutrophil count (ANC) ≥ 1,500/mm3.
* Platelet count ≥ 100,000/mm3.
* Total bilirubin within normal limits, 0-1 mg/dL.
* AST and ALT< 1.5 times ULN. (For patients with liver involvement: AST and ALT≤ 2.5 ULN).
* International normalized ratio (INR) < 2, prothrombin time (PT) < 20 sec, and partial thromboplastin time (PTT) < 55 sec .
* Creatinine < 1.5 x the ULN or GFR<45 ml/min.

Exclusion Criteria:

* HER-2 positive esophagogastric cancer. Patients with unknown HER2 status are permitted.
* Patients receiving any concurrent anticancer therapy or investigational agents with the intention of treating esophagogastric cancer. Last prior therapy must have been completed at least 2 weeks (14 days) prior to starting Nintedanib.
* Concurrent radiotherapy is not permitted for disease progression on treatment on protocol. However, symptomatic treatment for pre-existing non-target lesions would be allowed with approval from the principal investigator.
* Prior treatment with VEGFR inhibitor.
* Brain metastases or leptomeningeal disease.
* History of arterial thromboembolic (arterial blood clot) or hemorrhagic event with the exception of patients with pulmonary embolism stable on an anticoagulation regimen.
* Patients with a cerebrovascular accident or transient ischemic attack within the past six months.
* Patients on warfarin for any reason.
* Patient with known pre-existing interstitial lung disease.
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure, New York Heart Association (NYHA) functional classification of 3, unstable angina or poorly controlled arrhythmia. Myocardial infarction within 6 month prior to the study entry.
* Patients with history of proteinuria grade ≥ 2.
* Women of childbearing potential (WOCBP), or men who are able to father a child, unwilling to use a medically acceptable method of contraception during the trial and for at least three months after the end of active therapy.
* Women who are pregnant or breast-feeding. Persistence of clinically relevant therapy related toxicity from previous chemotherapy and/or radiotherapy. This does not include hemoglobin or other hematologic or laboratory criteria, as long as eligibility criteria are met
* Other malignancies within the past 5 years other than non-melanoma superficial skin cancer or carcinoma in situ of the cervix.
* Concurrent medical conditions or injury which may increase the risk of toxicity, including ongoing or active infection, history of significant bleeding disorder unrelated to cancer (congenital bleeding disorders, acquired bleeding disorders within one year), history of HIV-positive, or active or chronic hepatitis C and/or B infection.
* Known or suspected active drug or alcohol abuse.
* Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug. Patients who are unable to orally swallow the study medication.
* Known hypersensitivity to trial drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-09-04 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Janjigian, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center 1275 York Avenue, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nintedanib
Started | 34
Completed | 32
Not Completed | 2
Not completed — Participant not treated | 2

BASELINE CHARACTERISTICS:
Arm/Group | Nintedanib
Number analyzed (Participants) | 34
Age, Customized [Median (Full Range); unit: years] | 60 [34 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 28
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression-free Survival (PFS)
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nintedanib
Number analyzed (Participants) | 32
months | 1.9 [1.6 to 3.6]

2. Secondary Outcome: Objective Response Rate
Description: defined as both complete response (CR) and partial response (PR), as measured by RECIST response criteria.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib
Number analyzed (Participants) | 32
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 14
  Progressive Disease | 18

3. Secondary Outcome: Participants Evaluated for Toxicities
Description: The severity of adverse event should be classified and recorded according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib
Number analyzed (Participants) | 32
Participants | 32

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Nintedanib
All-Cause Mortality (participants affected / at risk) | 26/34
Serious Adverse Events (participants affected / at risk) | 8/34
Other Adverse Events (participants affected / at risk) | 32/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=34)
Anemia (Blood and lymphatic system disorders) | 1
Heart Failure (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 3
Fatigue (General disorders) | 2
Fever (General disorders) | 1
Skin infection (Infections and infestations) | 1
Blood bilirubin increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Skin & subcutaneous tissue disorders, Other, spec (Skin and subcutaneous tissue disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=34)
Fatigue (General disorders) | 18
Hypertension (Vascular disorders) | 16
Diarrhea (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 13
Aspartate aminotransferase increased (Investigations) | 12
Alanine aminotransferase increased (Investigations) | 11
Alkaline phosphatase increased (Investigations) | 11
Platelet count decreased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
White blood cell decreased (Investigations) | 4
Anemia (Blood and lymphatic system disorders) | 3
Blood bilirubin increased (Investigations) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Lymphocyte count decreased (Investigations) | 2
Mucositis oral (Gastrointestinal disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT02234596/Prot_SAP_000.pdf